CLINICAL TRIAL: NCT06864611
Title: Evaluating Huddles As a Novel Approach to Improving Concussion Safety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Kroshus, Research Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD114797-01A1 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: concussion; brain injury; prevention
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- US Soccer concussion education as usual. (No Intervention): Currently, US Soccer makes web-based concussion education information available, including a video about concussion reporting called "Recognize to Recover."
- Pre-Game Safety Huddles (Experimental)
  Interventions: Behavioral: Pre-Game Safety Huddles

INTERVENTIONS:
Behavioral: Pre-Game Safety Huddles — Before every regular season game, participating teams in league randomized to the Pre-Game Safety Huddle condition will hold brief Pre-Game Safety Huddles. Pre-Game Safety Huddles have three core components: (1) Gather (Athletes, coaches, officials, and other stakeholders come together before the start of the game); (2) Share (Opinion leaders (coaches, referees) affirm the importance of seeking care for suspected concussion, and (3) Repeat (Process is repeated before every game)
  Arms: Pre-Game Safety Huddles

SUMMARY:
Investigators will conduct a randomized controlled trial assessing the effectiveness and implementations of Pre-Game Safety Huddles (Huddles) in youth soccer.

DETAILED DESCRIPTION:
The clinical trial portion of this study will enroll 16 youth soccer leagues within four US states. Within each participating league we will enroll two "brackets" (closed units of teams at the same level that compete against each other during the regular season of play) of U12 boys' and girls' U12 teams. Based on typical league and bracket size we anticipate will be 384 teams. Randomization will happen at the league-level. Leagues in the Huddle intervention condition will be supported by US Soccer in implementing Pre-Game Safety Huddles before each regular season game. Leagues in the control condition will continue US Soccer's standard concussion education prevention activities.

Our primary effectiveness and implementation outcomes will be measured at the end of the regular season of play (anticipated to be 10 weeks). Maintenance outcomes will be measured at the end of the regular season of play one year later.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 9 and 13 on eligible teams in participating leagues.
* Soccer coaches of children between the ages of 9 and 13 on eligible teams in participating leagues.
* Read and write English

Exclusion Criteria:

* Cannot read and write English

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Expected concussion reporting behavior (Concussion Reporting- Expectations scale) | Baseline, 10 weeks (end of regular competitive season)
  Concussion Reporting- Expectations (CR-E), a 4-item scale that assesses athlete's expectations that they would tell a coach or other trusted adult about post-impact concussive symptoms in naturalistic scenarios. Responses are measured on a 4-point Likert scale, with higher sores indicating a stronger expectation that they would report future post-impact concussive symptoms.
Identification of suspected concussions | Baseline, 10 weeks (end of regular competitive season)
  Identification of suspected concussions will be measured via coach report as the number of times per season an athlete was identified as having a possible concussion (from 1- athlete-report to a coach, medical personnel or parent report to a coach, or 2- athlete removal from play for suspected concussive symptoms without report, for example due to loss of consciousness). This will be expressed as a team-level rate (number of instances/number of athletes per team).

SECONDARY OUTCOMES:
Perceived concussion reporting norms - Athlete (CR-N) | Baseline, 10 weeks (end of regular competitive season)
  CR-N is a 4-item scale that assesses the coach's perception that coaches in their organization would want athletes to report suspected concussive symptoms. Responses to four scenarios are measured on a 4-point Likert scale, with higher sores indicating a stronger perceived norms in support of reporting future post-impact concussive symptoms.
Perceived concussion reporting norms - Coach (CR-N) | Baseline, 10 weeks (end of regular competitive season)
  CR-N is a 4-item scale that assesses the coach's perception that coaches in their organization would want athletes to report suspected concussive symptoms. Responses to four scenarios are measured on a 4-point Likert scale, with higher sores indicating a stronger perceived norms in support of reporting future post-impact concussive symptoms.
Huddle implementation | 10 weeks (end of regular competitive season), 1 year and 10 weeks (end of following year's regular competitive season)
  Administrative data will be used to record the number of games before which Huddles occurred, which will be expressed as a rate with a denominator of Huddle-eligible games.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kroshus, Principal Investigator — Seattle Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in a publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.